CLINICAL TRIAL: NCT01690923
Title: Nasal Pillows at High CPAP Pressure
Brief Title: Nasal Pillows vs. Nasal Masks at High CPAP Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MA000-1442
Record Dates: First submitted 2012-09-16; First posted 2012-09-24 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-09

CONDITIONS: OSA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasal Mask First, then Pillows Mask (Experimental): Nasal mask is used for 7 nights, then followed by Pillows mask for 7 nights.
  [Nasal mask=Mirage Activa, Micro, FX; Pillows mask=Swift FX]
  Interventions: Device: Nasal mask; Device: Pillows mask
- Pillows Mask, then Nasal Mask (Experimental): Pillows mask for 7 nights, then followed by Nasal mask is used for 7 nights. [Nasal mask=MMirage Activa, Micro, FX; Pillows mask=Swift FX]
  Interventions: Device: Nasal mask; Device: Pillows mask

INTERVENTIONS:
Device: Nasal mask — Nasal mask (Mirage Activa, Micro, FX)
Device: Pillows mask — Nasal pillows mask (Swift FX)

SUMMARY:
The aim of this evaluation is to test:

1. Whether using nasal pillows at high pressures has comparable outcomes to nasal masks
2. Patient mask type preferences at high pressures

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to give written informed consent
* Patients who can read and comprehend English
* Patients being treated for OSA for >6 months
* Patients ≥ 18 years of age
* Patients using nasal mask systems with fixed pressure ≥ 12 cm H2O
* Patients who can trial the trial masks up to 14 nights
* Patients naive to pillows mask systems

Exclusion Criteria:

* Patients using an inappropriate mask system
* Patients using Bilevel flow generators
* Patients who are pregnant
* Patients who have a pre-existing lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schindhelm, Prof, Principal Investigator — ResMed
Locations (1):
- ResMed, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Zhu X, Wimms AJ, Benjafield AV. Assessment of the performance of nasal pillows at high CPAP pressures. J Clin Sleep Med. 2013 Sep 15;9(9):873-7. doi: 10.5664/jcsm.2984. PMID 23997699

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from ResMed Science Centre, Sydney, between Aug 2011 and Aug 2012
Groups:
- Nasal Mask First, Then Pillows Mask: Sequence 1: Nasal mask first, then Pillows mask
  [Nasal mask : Nasal mask (Mirage Activa, Micro, FX) Pillows mask : Nasal pillows mask (Swift FX)]
- Pillows Mask First, Then Nasal Mask: Sequence 2: Pillows mask first, then Nasal mask
  [Nasal mask : Nasal mask (Mirage Activa, Micro, FX) Pillows mask : Nasal pillows mask (Swift FX)]
Period: Overall Study
Arm/Group | Nasal Mask First, Then Pillows Mask | Pillows Mask First, Then Nasal Mask
Started | 10 | 11 (1 participant was withdrawn and excluded due to poor fit with the pillows mask)
Completed | 10 | 10
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Current CPAP Users: Nasal mask; Pillows mask
  Nasal mask : Nasal mask (Mirage Activa, Micro, FX)
  Pillows mask : Nasal pillows mask (Swift FX)
Arm/Group | Current CPAP Users
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Region of Enrollment [Number; unit: participants]
  Australia | 20

OUTCOME MEASURES:

1. Secondary Outcome: Usability
Description: Participant's feedback of performance of the study devices. Likert Scale 0-10 (0=very bad, 10=very good)
Time Frame: After 7 days of use
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Current CPAP Users
Number analyzed (Participants) | 20
Units on a scale
  Subjective Scores Overall Performance-Nasal Mask | 8.0 [7.25 to 9.75]
  Subjective Scores Overall Performance-Nasal Pillow | 8.5 [7 to 9]

2. Primary Outcome: AHI on Nasal Mask and Pillows Mask
Description: AHI (measure of sleep-disordered breathing severity) on nasal mask and nasal pillows measured as average events/hour
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Current CPAP Users
Number analyzed (Participants) | 20
events/hour
  AHI on nasal mask | 1.7 (1.1)
  AHI on Nasal pillows | 1.9 (1.3)

ADVERSE EVENTS:
Time Frame: 14 days
Description: Adverse events were collected for the study participation period of 14 days. Adverse events were collected/ assessed through clinical interview. No adverse events were reported or observed during the study.
Arm/Group | Current CPAP Users
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
This study only included established CPAP users.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No